CLINICAL TRIAL: NCT01982045
Title: A Randomized Controlled Trial of AttraX® Putty vs. Autograft in Instrumented Posterolateral Spinal Fusion
Brief Title: RCT of AttraX® Putty vs. Autograft in Instrumented Posterolateral Spinal Fusion
Acronym: AxA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: NuVasive (Industry)
Responsible Party: Principal Investigator, M.C. Kruyt, MD, PhD, Orthopaedic surgeon, UMC Utrecht
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NL44095.041.13
Record Dates: First submitted 2013-10-28; First posted 2013-11-13 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Spinal Deformity; Spinal Instability; Instrumented Spinal Fusion
Keywords: Bone graft; Ceramic; Spinal fusion; RCT; Thoracolumbar region

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AttraX condition (Experimental): 8-10cc of AttraX® Putty per spinal level at the randomized allocation side of the spine (left or right).
  Interventions: Device: AttraX® Putty
- Autograft condition (Active Comparator): 8-10cc autologous bone graft per spinal level at the control side of the spine. This can be a combination of local bone and iliac crest bone, but at least 50% of the volume has to be iliac crest bone graft.
  Interventions: Other: Autologous bone graft

INTERVENTIONS:
Device: AttraX® Putty — Synthetic bone graft comprised of calcium phosphate granules and hydroxyapatite with an advanced biodissolvable polymer carrier that allows for better handling of the granules in putty form.
  Arms: AttraX condition
Other: Autologous bone graft — Corticocancellous bone harvested from the iliac crest, with our without local bone obtained from decompression and/or preparation for fusion (facetectomy and denudement).
  Arms: Autograft condition

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of AttraX® Putty as a bone graft substitute for autograft in instrumented posterolateral fusion of the thoracolumbar spine, in terms of efficacy and safety.

DETAILED DESCRIPTION:
Spinal fusion, a surgical procedure frequently used for many spinal conditions requiring stabilization of the vertebral column, is currently performed by using large amounts of autologous bone graft or autograft. A substitute for this patient own bone would eliminate the graft harvesting morbidity that is currently one of the main disadvantages. Recently, a promising synthetic graft substitute has been developed that has shown favorable results in pre-clinical studies. This product is AttraX® Putty (CE-557130), a bioresorbable tricalcium phosphate (TCP), mixed with a fast resorbing polymer carrier to improve surgical handling. The aim of the current study is to clinically investigate AttraX® Putty as an alternative to autologous bone graft in adult patients qualified for instrumented posterolateral fusion of the thoracolumbar spine (T10-S1).

The study design is a patient and observer blinded, controlled, randomized, multi-center clinical trial with intra-patient comparisons. This means that each patient is it owns control. According to a randomization scheme, one side of the spine will be grafted with AttraX® Putty the other side receives bone harvest from the iliac crest, which is currently the gold standard.

The primary outcomes of this study are the posterior spinal fusion rate after one year (based on CT-scans), and potential serious adverse events related with AttraX® Putty. Secondary outcomes are the resorption characteristics during the first year, volume of bridging bone mass after one year, evaluation of iliac crest pain, correlation of the posterior fusion rate to the presence of interbody fusion after one year and the posterior spinal fusion rate after two years.

ELIGIBILITY:
Inclusion Criteria:

* To be treated with instrumented posterolateral thoracolumbar spinal fusion, with or without additional posteriorly inserted interbody devices (PLIF, TLIF), because of (1) deformity, (2) structural instability and/or (3) expected instability as a result of decompression for spinal stenosis;
* Non-responsive to at least 6 months of non-operative treatment prior to study enrollment;
* Fusion indicated for one or more levels in the T10 to S1/ilium region;
* Willing and able to understand and sign the study specific Patient Informed Consent;
* Skeletally mature between 18 and 80 years of age;

Exclusion Criteria:

* Any previous surgical attempt(s) for spinal fusion (revision surgery);
* Previous treatments that compromise fusion surgery like irradiation;
* Previous autologous bone grafting procedures that compromise the quality and amount of iliac crest bone grafting;
* Indication for spinal fusion because of a traumatic reason, like a spinal fracture or traumatic instability;
* Active spinal and/or systemic infection;
* Spinal metastasis in the area intended for fusion;
* Systemic disease or condition, which would affect the subjects ability to participate in the study requirements or the ability to evaluate the efficacy of the graft (e.g. active malignancy, neuropathy);
* At risk to be non-compliant (e.g. (recently treated for) substance abuse, detainee, likely to immigrate);
* Participation in clinical trials evaluating investigational devices, pharmaceuticals or biologics within 3 months of enrollment in the study;
* Female patients who intend to be pregnant within 1.5 year of enrollment in the study;
* Body mass index (BMI) larger than 35 (morbidly obese);
* Being expected to require additional surgery to the same spinal region within the next 6 months;
* Current or recent (<1yr) corticosteroid use equivalent to prednisone ≥5mg/day, prescribed for more than 6 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Posterior spinal fusion rate after one year | One year (12-15 months) after surgery
  For the efficacy analysis of AttraX® Putty as a bone graft substitute for autograft in instrumented posterolateral fusion of the thoracolumbar spine, a comparison will be made between the fusion performance of the AttraX condition and the autograft condition after one year, assessed at CT-scans. Non-inferiority of AttraX® Putty will be tested with a McNemar's test.
Rate of (serious) adverse events with a potential relation with AttraX® Putty | Untill 2 years (24-27 months) after surgery
  The safety of AttraX® Putty will be evaluated by documenting the number and nature of all (serious) adverse events that occur within the study population. The complication rate will be compared to the rate in control populations from the UMC Utrecht and a recently performed comparable multicenter-RCT coordinated by the UMC Utrecht. In addition, all (serious) adverse events will be evaluated for any potential relation with AttraX® Putty.

SECONDARY OUTCOMES:
Resorption characteristics of AttraX® Putty compared to autograft during the first year | During the first year (12-15 months) after surgery
  In a subset of the study population, additional DEXA-scans at 1-5 days after surgery (reference scan) and at 6 weeks, 3 months, 6 months and 1 year follow-up will be made to evaluate the resorption characteristics of AttraX® Putty compared to autograft in the instrumented fusion locations.
Volume of bridging bone mass after one year | One year (12-15 months) after surgery
  As quantification of the bone mass volume allows more detailed investigation of the amount of bone that has been formed, the volume of bridging bone mass derived from AttraX® Putty will be compared with the bone mass derived from autograft, using the one year CT scans made for the primary objective.
Visual analogue pain scale of iliac crest pain | During two years (24-27 months) after surgery
  Assessments of iliac crest pain at 6 weeks, 3 months, 6 months, 1 year and 2 years follow-up, by patients blinded to the side of graft harvesting from the iliac crest, will be analysed to investigate the relevance of donor site pain.
Correlation of posterior fusion rate to the presence of interbody fusion after one year | One year (12-15 months) after surgery
  The correlation of the posterior fusion rate to the presence of interbody fusion will be assessed at the one year CT scans made for the primary objective.
Posterior spinal fusion rate after two years | Two years (24-27 months) after surgery
  To determine the long-term fusion potential and behavior from AttraX® Putty and autograft, a comparison will be made between the fusion performance of both conditions after two years, assessed at CT-scans. Only those patients that scored a doubtful fusion or non-union in any of the relevant levels at the one-year CT scan will be scanned.

CONTACTS AND LOCATIONS:
Overall Officials: Moyo Kruyt, MD, PhD, Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Lehr AM, Jacobs WC, Stellato RK, Castelein RM, Cumhur Oner F, Kruyt MC. Methodological aspects of a randomized within-patient concurrent controlled design for clinical trials in spine surgery. Clin Trials. 2022 Jun;19(3):259-266. doi: 10.1177/17407745221084705. Epub 2022 Mar 17. PMID 35297288